CLINICAL TRIAL: NCT02530424
Title: "Neo-Adjuvant Treatment With the CDK4,6 Inhibitor Palbociclib in HER2-positive and ER-positive Breast Cancer: Effect on Ki67 and Apoptosis Before, During and After Treatment "
Brief Title: "Neo-Adjuvant Treatment With Palbociclib: Effect on Ki67 and Apoptosis Before, During and After Treatment "
Acronym: NA-PHER2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Michelangelo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FM-14-B01
Record Dates: First submitted 2014-09-19; First posted 2015-08-21 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2019-07

CONDITIONS: Breast Neoplasms
Keywords: HER2-positive; ER-positive; invasive; CDK4,6; Palbociclib; neoadjuvant treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; pertuzumab; palbociclib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trast-pert-palbo-fulve (Experimental): Patients will receive an association of drugs (trastuzumab, pertuzumab, palbociclib plus or minus fulvestrant) as neoadjuvant chemotherapy. Definitive surgery will be performed not earlier than 14 days and not later than 28 days after the last dose of any of the drugs in the combination. After completion of surgical treatment patients will receive irradiation as locally acceptable.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Palbociclib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab (8 mg/kg loading dose IV, then 6 mg/kg IV) will be given on day 1 q. 3 weeks for a total of 6 administrations
  Other Names: Herceptin
Drug: Pertuzumab — Pertuzumab (840 mg as an i.v. infusion) will be given on day 1 q. 3 weeks for a total of 6 administration
  Other Names: Perjeta
Drug: Palbociclib — Palbociclib will be given at the dose of 125 mg po q.d. x 21 every 4 weeks (i.e. 1 week rest period for a total of 5 cycles
  Other Names: Ibrabce
Drug: Fulvestrant — Fulvestrant will be administered according to local prescription guidelines and will be given intra-muscle at the dose of 500 mg every 4 weeks (repeat for 5 times) with an additional 500 mg dose given two weeks after the initial dose
  Other Names: Faslodex

SUMMARY:
This is a multicenter neoadjuvant trial conducted under the sponsorship and overall trial management of the Fondazione Michelangelo in Italy.

Women with a diagnosis of invasive unilateral non metastatic ER-positive breast cancer expressing HER2 and suitable for neoadjuvant therapy Patients in this study will receive: Trastuzumab+Pertuzumab+Palbociclib with or without Fulvestrant (HPPF)

Trastuzumab 8 mg/kg loading dose IV, then 6 mg/kg IV q.3 wks (repeat for a total of 6 administrations) Pertuzumab 840 mg loading dose IV, then 420 mg IV q. 3 wks (repeat for a total of 6 administrations) Palbociclib 125 mg po q.d. x 21 q. 4 wks (= 1 cycle; repeat for a total of 5 cycles) Fulvestrant will be given intra-muscle at the dose of 500 mg every 4 weeks (repeat for 5 times) with an additional 500 mg dose given two weeks after the initial dose (total administrations including the additional one = 6)

The total duration of neoadjuvant palbociclib (5 cycles every 4 weeks) and fulvestrant (5 administrations every 4 weeks plus the additional dose given two weeks after the initial dose) was selected to match as closely as possible the total duration of the six planned 3-weekly administrations of trastuzumab and pertuzumab

Definitive surgery will be performed not earlier than 14 days and not later than 28 days after the last dose of any of the drugs in the combination reported above

After completion of the neoadjuvant and surgical treatment patients will receive irradiation as locally acceptable.

Patients will also continue to receive systemic drug therapy including chemotherapy (plus standard anti-HER2 treatment until completion of full 1 year if HER2 3+ or neu amplified, i.e. cohorts A and B) and endocrine therapy according to local guidelines at the Investigator's discretion.

DETAILED DESCRIPTION:
This is a multicenter neoadjuvant trial conducted under the sponsorship and overall trial management of the Fondazione Michelangelo in Italy.

Three cohorts of patients are planned

Patients with ER positive tumors (> 10%) and HER2 3+ or neu amplified Cohort A Trastuzumab+Pertuzumab+Palbociclib+Fulvestrant (HPPF)

Cohort B Trastuzumab+Pertuzumab+Palbociclib (HPP) Allocation to Cohort B will be started after recruitment to Cohort A has been completed

Patients with ER positive tumors (> 10%), PgR positive, HER2 1+/2+ (without amplification) and Ki67 > 20% Cohort C Trastuzumab+Pertuzumab+Palbociclib+Fulvestrant (HPPF)

Trastuzumab 8 mg/kg loading dose IV, then 6 mg/kg IV q.3 wks (repeat for a total of 6 administrations) Pertuzumab 840 mg loading dose IV, then 420 mg IV q. 3 wks (repeat for a total of 6 administrations) Palbociclib 125 mg po q.d. x 21 q. 4 wks (= 1 cycle; repeat for a total of 5 cycles) Fulvestrant will be given intra-muscle at the dose of 500 mg every 4 weeks (repeat for 5 times) with an additional 500 mg dose given two weeks after the initial dose (total administrations including the additional one = 6)

The total duration of neoadjuvant palbociclib (5 cycles every 4 weeks) and fulvestrant (5 administrations every 4 weeks plus the additional dose given two weeks after the initial dose) was selected to match as closely as possible the total duration of the six planned 3-weekly administrations of trastuzumab and pertuzumab

Definitive surgery will be performed not earlier than 14 days and not later than 28 days after the last dose of any of the drugs in the combination reported above

After completion of the neoadjuvant and surgical treatment patients will receive irradiation as locally acceptable.

Patients will also continue to receive systemic drug therapy including chemotherapy (plus standard anti-HER2 treatment until completion of full 1 year if HER2 3+ or neu amplified, i.e. cohorts A and B) and endocrine therapy according to local guidelines at the Investigator's discretion.

Primary objectives:

* Characterize changes of Ki67 from baseline before therapy and at 2 weeks and at surgery (approximately 22 weeks after start of neoadjuvant therapy with HPPF).
* Characterize changes in apoptosis from baseline before therapy and at surgery (approximately 22 weeks after start of neoadjuvant therapy with HPPF).
* Study the tolerability profile of the combination

Secondary objectives:

* Assess the rate of pathological complete response (pCR) defined as ypT0-ypTis ypN0 at surgery
* Define the clinical objective response rate at the end of the combination
* Conduct molecular and clinical analyses to assess the presence of informative markers of benefit in addition to Ki67 and apoptosis

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18 years or older with tumors suitable for neoadjuvant treatment
2. Early (> 1.5 cm) or locally advanced untreated breast cancer
3. Histologically confirmed invasive unilateral breast cancer
4. HER2 status to be centrally confirmed (HER2 3+ of neu amplified for cohorts A and B; HER2 1+/2+ without amplification for cohort C)
5. Positive estrogen receptor (ER) > 10% and known progesterone receptor (PgR). Note: PgR assessment must be positive for cohort C
6. Ki67 > 20% for cohort C
7. Available paraffin-embedded tumor block taken at diagnostic biopsy for central retrospective confirmation of HER2 and ER eligibility and for assessment of Ki67 value and apoptosis is mandatory
8. All patients must agree to provide tumor tissues for centralized assessment of KI67 values and apoptosis at the required timelines (2 weeks from starting protocol therapy and at surgery)
9. ECOG (Eastern Cooperative Oncology Group) performance status 0 or 1
10. Written informed consent to participate in the trial (approved by the Institutional Review Board/ Independent Ethics Committee) obtained prior to any study specific screening procedures
11. Willing and able to comply with the protocol

Exclusion Criteria:

1. Evidence of bilateral invasive breast cancer or metastatic disease (M1)
2. Pregnant or lactating women.
3. Women with childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception
4. Previous treatment with chemotherapy, hormonal therapy or an investigational drug for any type of malignancy
5. Previous extensive radiotherapy
6. Previous investigational treatment for any condition within 4 weeks of registration date
7. Known hypersensitivity reaction to one of the compounds or incorporated substances used in this protocol
8. Previous or concomitant malignancy of any other type that could affect compliance with the protocol or interpretation of results.
9. Other serious illness or medical condition including: history of documented congestive cardiac failure; angina pectoris requiring anti-anginal medication; evidence of transmural infarction on ECG; poorly controlled hypertension; clinically significant valvular heart disease; high-risk uncontrolled arrhythmias
10. Baseline left ventricular ejection fraction (LVEF) < 55% by echocardiography or multi-gated scintigraphic scan (MUGA)
11. QTc (corrected QT interval) >480 msec or a family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes (TdP)
12. Patients with a history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant and precluding informed consent or adversely affecting compliance with study drugs
13. Serious uncontrolled infections (bacterial or viral) or poorly controlled diabetes mellitus
14. Current use or anticipated need for food or drugs that are known strong CYP3A4 (cytochrome P450 3A4) inhibitors or inducers
15. Uncontrolled electrolyte disorders that can compound the effects of a QTc prolonging drug (e.g., hypocalcemia, hypokalemia, hypomagnesemia)
16. Abnormal baseline hematological values:
17. Abnormal baseline liver function, bilirubin, creatinine and/or INR (international normalized ratio)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-05; Primary Completion 2019-09 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Serial measures of Ki67 | Participants will be followed for the duration of protocol therapy, an expected average of 26 weeks
  Changes in Ki67 scores from baseline before therapy, 2 weeks after and then at surgery
Serial measures of apoptosis | Participants will be followed for the duration of protocol therapy, an expected average of 26 weeks
  Changes in apoptosis biomarker scores from baseline before therapy and at surgery

SECONDARY OUTCOMES:
pathological complete response (pCR) | at surgery
  Assess the rate of pathological complete response (pCR) defined as ypT0-ypTis ypN0 at surgery
clinical objective response | Participants will be followed for the duration of medical therapy, an expected average of 24 weeks
  Assess the clinical objective response rate after medical therapy
Number of participants with adverse events as a Measure of Safety and Tolerability | Participants will be followed for up to 7 months
  Number of participants with Adverse Events and related grade

CONTACTS AND LOCATIONS:
Overall Officials: Luca Gianni, MD, Study Chair — Ospedale San Raffaele
Locations (7):
- Italy (7):
  - Policlinico Sant'Orsola Malpighi, Bologna, BO
  - Azienda Ospedaliero Universitaria di Ferrara - Arcispedale S. Anna, Ferrara, FE
  - IST San Martino, Genova, GE
  - Ospedale San Raffaele, Milan, MI
  - Istituto Europeo di Oncologia, Milan, MI
  - Arcispedale S.Maria Nuova A.O.Reggio Emilia, Reggio Emilia, RE
  - Ospedale Santa Maria della Misericordia, Udine, UD

REFERENCES:
- [Derived] Vigano L, Locatelli A, Ulisse A, Galbardi B, Dugo M, Tosi D, Tacchetti C, Daniele T, Gyorffy B, Sica L, Macchini M, Zambetti M, Zambelli S, Bianchini G, Gianni L. Modulation of the Estrogen/erbB2 Receptors Cross-talk by CDK4/6 Inhibition Triggers Sustained Senescence in Estrogen Receptor- and ErbB2-positive Breast Cancer. Clin Cancer Res. 2022 May 13;28(10):2167-2179. doi: 10.1158/1078-0432.CCR-21-3185. PMID 35254385
- [Derived] Gianni L, Colleoni M, Bisagni G, Mansutti M, Zamagni C, Del Mastro L, Zambelli S, Bianchini G, Frassoldati A, Maffeis I, Valagussa P, Viale G. Effects of neoadjuvant trastuzumab, pertuzumab and palbociclib on Ki67 in HER2 and ER-positive breast cancer. NPJ Breast Cancer. 2022 Jan 10;8(1):1. doi: 10.1038/s41523-021-00377-8. PMID 35013314
- [Derived] Gianni L, Bisagni G, Colleoni M, Del Mastro L, Zamagni C, Mansutti M, Zambetti M, Frassoldati A, De Fato R, Valagussa P, Viale G. Neoadjuvant treatment with trastuzumab and pertuzumab plus palbociclib and fulvestrant in HER2-positive, ER-positive breast cancer (NA-PHER2): an exploratory, open-label, phase 2 study. Lancet Oncol. 2018 Feb;19(2):249-256. doi: 10.1016/S1470-2045(18)30001-9. Epub 2018 Jan 8. PMID 29326029